CLINICAL TRIAL: NCT00724399
Title: Preventive Health Practices in Women
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ruth Carlos M.D., Primary Investigator, University of Michigan
Other Study IDs: HUM00010173
Record Dates: First submitted 2008-07-24; First posted 2008-07-29 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Observations: Women attending screening mammography and gynecology visit
  Interventions: Behavioral: Survey on womens health Issues.
- A: Women attending their annual screening mammography and gynecology clinic visits.

INTERVENTIONS:
Behavioral: Survey on womens health Issues. — Cardiovascular health.
  Groups: Observations

SUMMARY:
The purpose of this study is to evaluate women's level of knowledge and health practices regarding cardiovascular health and identify barriers to appropriate health practice.

DETAILED DESCRIPTION:
Increasingly, gender differences in manifestation of cardiovascular disease (CVD) and myocardial infarction (MI) are being reported. Gender specific presentations of MI in particular have contributed to underdiagnosis of cardiac events in women. Furthermore, previous studies from the 2002 Behavioral Risk Factors Screening Surveillance demonstrated decreased compliance with standard cardiovascular health practices in women compared to men. We seek to validate these findings in a population of women undergoing screening mammography and annual gynecology visit to identify current state of knowledge regarding cardiovascular risk in women.

ELIGIBILITY:
Inclusion Criteria:

* Women attending screening mammography and gynecology visit.

Exclusion Criteria:

* Patient refusal to participate (assessed by non-submission of the completed survey).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prospective survey study on women who attend screening mammography and routine/annual gynecology visits to assess baseline knowledge regarding CVD.
Sampling Method: Non-Probability Sample
Enrollment: 1418 (Actual)
Dates: Start 2006-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To validate findings in a population of women undergoing screening mammography and annual gynecology visit to identify current state of knowledge regarding cardiovascular risk in women. | To be determined later

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Carlos, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No